CLINICAL TRIAL: NCT05627180
Title: Tailored Health Literacy Follow-up in Cancer - the Tail HealthLit Cancer Trial
Brief Title: Tailored Health Literacy Follow-up in Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Christine Råheim Borge, Researcher, Lovisenberg Diakonale Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 341
Record Dates: First submitted 2022-11-10; First posted 2022-11-25 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Cancer
Keywords: Health literacy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator
Masking Description: The main researcher and PhD candidate will be blinded to the randomizing procedure. However, in this project, it is not feasible to blind the participants, HCPs or PhD candidate to the participants' group. The participants will be randomized right after the first assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Intervention Group (Experimental): The intervention group will receive a tailored intervention based on each individuals health literacy needs. A project nurse with broad experience in cancer care will be trained in Motivational Interviewing techniques to provide follow-up for the patients in the intervention group in a period of 9 months.
  Interventions: Behavioral: Tailored Health Literacy follow-up in cancer
- Usual care group (No Intervention): Usual care group will receive usual follow-up.

INTERVENTIONS:
Behavioral: Tailored Health Literacy follow-up in cancer — 1. Participants are invited to a consultation with the project nurse where the project nurse will use baseline data to identify the patient's HL needs, QOL, symptom burden and issues related to self-management of their cancer and treatment. These data will be used together with an interview questionnaire specifically developed to communicate HL needs (i.e. CHAT), which form the basis for the individualized HL support.
  2. Actions: Based on results of the consultation, the project nurse and the patient will use a worksheet of possible actions to identify those most relevant to the patient's individual needs. Based on this, different self-management tasks and actions will be offered, and an individual tailored follow-up plan will be made. The patient and the project nurse will use a workbook containing information on the follow-up plan that will be added into medical record.
  3. Telephone/digital conversations with the project every second month for a period of 9 months.
  Arms: The Intervention Group

SUMMARY:
Health literacy refers to personal and relational factors affecting a persons ability to aquire, understand and use health information and health services. In a need assessment study, it was found that there is a need to focus on health literacy factors in the follow-up of people with cancer in the health care services.

Thus, this project evaluate the effect of a health literacy intervention in cancer. The intervention provides patients with nurse-led tailored follow-up by phone/digital/personal meetings that addresses their individual HL needs, particularly those needs that impact their quality of life, symptom burden, self-management, and health economic costs. Our main goal is to improve the patients' health literacy, with secondary goals of improving their quality of life, symptom burden, and self-management, and reducing their health care costs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer
* Above 18 years old
* Receiving treatment at the main intervention hospital

Exclusion Criteria:

* Not diagnosed with cancer
* Not above 18 years old
* Not in treatment at the intervention hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
General Health literacy measured with the Health Literacy Questionnaire (HLQ) | 6 months, 9 months
  Change of Health Literacy questionnaire

SECONDARY OUTCOMES:
Electronic Health Literacy measured with the electronic Health Literacy Questionnaire (eHLQ) | 6 months, 9 months
  Change of electronic Health Literacy questionnaire
General symptoms measured with the Edmonton Symptom Assessment System (ESAS) | 6 months, 9 months
  Change of symptom burden questionnaire
Oral symptoms measured with four items selected from the European Organization for REsearch and Treatment of Cancer-oral health 15 (EORTC-OH 15) | 6 months, 9 months
  Change in oral symptoms
Self-management measured with the Health Education Impact Questionnaire (HeiQ) | 6 months, 9 months
  Change of self-management questionnaire
Self-Efficacy measured with the General Self-efficacy Scale (GSE) | 6 months, 9 months
  Change of Self-efficacy questionnaire
Disease specific Quality of Life measured with the The functional Assessment of Cancer Therapy-General (FACT-G) | 6 months, 9 months
  Change of quality of life questionnaire
Generic health-related quality of life/quality adjusted life years measured by the EQ-5D | 6 months, 9 months
  Change in health related quality of life and adjusted life years
Health care costs measured through collecting data from patient medical records, patient self-report, and data registers | 6 months, 9 months
  Change of health care costs

CONTACTS AND LOCATIONS:
Overall Officials: Christine R Borge, PhD, Principal Investigator — Lovisenberg Diaconal Hospital and University of Oslo; Astrid K Wahl, PhD, Study Chair — University of Oslo; Simen A Steindal, PhD, Study Chair — VID
Locations (1):
- Lovisenberg Diakonale Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No